CLINICAL TRIAL: NCT00576693
Title: Stenting vs. Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis
Acronym: SAMMPRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Marc Chimowitz, Full Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS058728-01A1; NINDS (Other: NINDS); CRC (Other: NINDS); 1U01NS058728-01A1 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-19 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; intracranial stenting; vascular risk factor management
MeSH Terms: conditions — Ischemic Stroke | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive medical management plus stenting (Experimental): intracranial angioplasty and stenting using the Gateway balloon and Wingspan self-expanding nitinol stent (or any future FDA approved iterations of the balloon, stent, or the delivery systems) plus intensive medical therapy (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl).
  Interventions: Device: intracranial angioplasty and stenting
- intensive medical management alone (Experimental): Intensive medical therapy alone (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl)
  Interventions: Other: intensive medical management

INTERVENTIONS:
Device: intracranial angioplasty and stenting — intracranial angioplasty and stenting using the Gateway balloon and Wingspan self-expanding nitinol stent (or any future FDA approved iterations of the balloon, stent, or the delivery systems) plus intensive medical therapy (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl).
  Other Names: Wingspan stent; Gateway balloon
  Arms: intensive medical management plus stenting
Other: intensive medical management — intensive medical therapy alone (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl)
  Arms: intensive medical management alone

SUMMARY:
PRIMARY HYPOTHESIS:

Compared with intensive medical therapy alone, intracranial angioplasty and stenting combined with intensive medical therapy will decrease the risk of the primary endpoint by 35% over a mean follow-up of two years in high-risk patients patients with 70% - 99% intracranial stenosis who had a transient ischemic attack (TIA) or stroke within 30 days prior to enrollment) with symptomatic stenosis of a major intracranial artery.

SUMMARY:

The best treatment for prevention of another stroke or TIA in patients with narrowing of one of the arteries in the brain is uncertain. A common treatment is the use of anti-clotting medications to prevent blood clots from forming in the narrowed vessel. There are a variety of medicines used for this purpose. These medications are usually taken for the rest of a patient's life.

However, a treatment that has been used successfully together with anti-clotting medications in patients with narrowing of the blood vessels of the heart is now being studied in the blood vessels of the brain. This treatment is called stenting.

Recent research has also indicated a benefit in prevention of recurring stroke by Intensive Medical Therapy, which is defined as treating risk factors for stroke like high blood pressure, elevated LDL (low density lipids - the "bad" form of cholesterol) and diabetes. The purpose of this study is to compare the safety and effectiveness of either Intensive Medical Therapy PLUS Stenting or Intensive Medical Therapy ONLY in preventing stroke, heart attacks or death.

The study will enroll patients over a 5 year period. Each participant will be involved in the study for a minimum of 1 year and a maximum of 3 years.

Fifty different medical centers in the United States are part of this study. Both the Clinical Coordinating Center and the Statistical Coordinating Center for the entire study will be located at Emory University.

DETAILED DESCRIPTION:
This will be an investigator initiated and designed Phase III multicenter trial in which patients with TIA or non-disabling stroke within 30 days prior to enrollment that is caused by 70% - 99% stenosis of a major intracranial artery (MCA, carotid, vertebral, or basilar) will be randomized (1:1) at approximately 50 sites to:

intensive medical therapy alone (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl)

OR

intracranial angioplasty and stenting using the Gateway balloon and Wingspan self-expanding nitinol stent (or any future FDA approved iterations of the balloon, stent, or the delivery systems) plus intensive medical therapy (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl).

Risk factor management will be performed by the study neurologist at each site who will be assisted by an innovative, evidence-based, educational, lifestyle modification program (INTERxVENT) that will be administered at regularly scheduled times to all patients throughout the study.

All patients enrolled in the trial will be followed until the first of the following: 90 days after a primary endpoint, death, or the close-out visit in the trial, which will occur within a window from 60 days before March 31, 2012 to 30 days after March 31, 2013. Patients who do not die or have a primary endpoint during follow-up will be followed for 2-4.5 years.

ELIGIBILITY:
INCLUSION CRITERIA

1. Transient ischemic attack (TIA) or non-severe stroke within 30 days of enrollment attributed to 70-99% stenosis of a major intracranial artery (carotid artery, MCA stem (M1), vertebral artery, or basilar artery)

   • may be diagnosed byTranscranial Doppler (TCD), Magnetic Resonance Angiogram (MRA), or computed tomography angiography (CTA) to qualify for angiogram performed as part of the study protocol but must be confirmed by catheter angiography for enrollment in the trial
2. Modified Rankin score of ≤ 3
3. Target area of stenosis in an intracranial artery that has a normal diameter of 2.00 mm to 4.50 mm
4. Target area of stenosis is less than or equal to 14 mm in length
5. Age ≥ 30 years and ≤ 80 years.

   • Patients 30-49 years are required to meet at least one additional criteria (i-vi) provided in the table below to qualify for the study. This additional requirement is to increase the likelihood that the symptomatic intracranial stenosis in patients 30-49 years is atherosclerotic.

   i. insulin dependent diabetes for at least 15 years ii. at least 2 of the following atherosclerotic risk factors: hypertension (BP > 140/90 or on antihypertensive therapy); dyslipidemia (LDL > 130 mg /dl or HDL < 40 mg/dl or fasting triglycerides > 150 mg/dl or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event ii. history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease iv. any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic v. aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography vi. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic
6. Negative pregnancy test in a female who has had any menses in the last 18 months
7. Patient is willing and able to return for all follow-up visits required by the protocol
8. Patient is available by phone
9. Patient understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent

EXCLUSION CRITERIA

1. Tandem extracranial or intracranial stenosis (70%-99%) or occlusion that is proximal or distal to the target intracranial lesion (NOTE: an exception is allowed if the occlusion involves a single vertebral artery proximal to a symptomatic basilar artery stenosis and the contralateral vertebral artery is supplying the basilar artery)
2. Bilateral intracranial vertebral artery stenosis of 70%-99% and uncertainty about which artery is symptomatic (e.g. if patient has pontine, midbrain, or temporal - occipital symptoms)
3. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to expected enrollment date
4. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform staged angioplasty followed by stenting of target lesion
5. Plan to perform concomitant angioplasty or stenting of an extracranial vessel tandem to an intracranial stenosis
6. Presence of intraluminal thrombus proximal to or at the target lesion
7. Any aneurysm proximal to or distal to stenotic intracranial artery
8. Intracranial tumor (except meningioma) or any intracranial vascular malformation
9. CT or angiographic evidence of severe calcification at target lesion
10. Thrombolytic therapy within 24 hours prior to enrollment
11. Progressive neurological signs within 24 hours prior to enrollment
12. Brain infarct within previous 30 days of enrollment that is of sufficient size (> 5 cms) to be at risk of hemorrhagic conversion during or after stenting
13. Any hemorrhagic infarct within 14 days prior to enrollment
14. Any hemorrhagic infarct within 15 - 30 days that is associated with mass effect
15. Any history of a primary intracerebral (parenchymal) hemorrhage (ICH)
16. Any other intracranial hemorrhage (subarachnoid, subdural, epidural) within 30 days
17. Any untreated chronic subdural hematoma of greater than 5 mm in thickness
18. Intracranial arterial stenosis due to arterial dissection, Moya Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with Cerebrospinal fluid (CSF) pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus
19. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%
20. Known allergy or contraindication to aspirin, clopidogrel, heparin, nitinol, local or general anesthesia
21. History of life-threatening allergy to contrast dye. If not life threatening and can be effectively pretreated, patient can be enrolled at physician's discretion
22. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets < 100,000, hematocrit < 30, International normalized ratio (INR) > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), severe liver impairment Aspartate Transaminase (AST) or Alanine transaminase (ALT) > 3 x normal, cirrhosis, creatinine > 3.0 (unless on dialysis)
23. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 90 days after enrollment
24. Indication for warfarin or heparin beyond enrollment (NOTE: exceptions allowed for use of systemic heparin during stenting procedure or subcutaneous heparin for deep vein thrombosis (DVT) prophylaxis while hospitalized)
25. Severe neurological deficit that renders the patient incapable of living independently
26. Dementia or psychiatric problem that prevents the patient from following an outpatient program reliably
27. Co-morbid conditions that may limit survival to less than 3 years
28. Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study
29. Enrollment in another study that would conflict with the current study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2008-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Chimowitz, MBChB, Principal Investigator — Medical University of South Carolina
Locations (50):
- United States (50):
  - UAB Medical Center, Birmingham, Alabama
  - Barrow Neurological Institute - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo, Phoenix, Arizona
  - Glendale Adventist, Glendale, California
  - Cedars Sinai, Los Angeles, California
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Washington Hospital, Washington D.C., District of Columbia
  - University of Florida - Shands, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State, Detroit, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Providence St. John, Southfield, Michigan
  - University of Mississippi, Jackson, Mississippi
  - University of Buffalo, Buffalo, New York
  - NYU Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses Cone Medical Center, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - Baylor St. Luke's, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Scott & White - Texas A&M, Temple, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentera, Norfolk, Virginia
  - Sacred Heart Medical Center, Spokane, Washington
  - MultiCare, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Derdeyn CP, Fiorella D, Lynn MJ, Barnwell SL, Zaidat OO, Meyers PM, Gobin YP, Dion J, Lane BF, Turan TN, Janis LS, Chimowitz MI; SAMMPRIS Trial Investigators. Impact of operator and site experience on outcomes after angioplasty and stenting in the SAMMPRIS trial. J Neurointerv Surg. 2013 Nov;5(6):528-33. doi: 10.1136/neurintsurg-2012-010504. Epub 2012 Sep 12. PMID 22977278
- [Result] Turan TN, Lynn MJ, Nizam A, Lane B, Egan BM, Le NA, Lopes-Virella MF, Hermayer KL, Benavente O, White CL, Brown WV, Caskey MF, Steiner MR, Vilardo N, Stufflebean A, Derdeyn CP, Fiorella D, Janis S, Chimowitz MI; SAMMPRIS Investigators. Rationale, design, and implementation of aggressive risk factor management in the Stenting and Aggressive Medical Management for Prevention of Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) trial. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):e51-60. doi: 10.1161/CIRCOUTCOMES.112.966911. No abstract available. PMID 22991350
- [Result] Fiorella D, Derdeyn CP, Lynn MJ, Barnwell SL, Hoh BL, Levy EI, Harrigan MR, Klucznik RP, McDougall CG, Pride GL Jr, Zaidat OO, Lutsep HL, Waters MF, Hourihane JM, Alexandrov AV, Chiu D, Clark JM, Johnson MD, Torbey MT, Rumboldt Z, Cloft HJ, Turan TN, Lane BF, Janis LS, Chimowitz MI; SAMMPRIS Trial Investigators. Detailed analysis of periprocedural strokes in patients undergoing intracranial stenting in Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS). Stroke. 2012 Oct;43(10):2682-8. doi: 10.1161/STROKEAHA.112.661173. Epub 2012 Sep 13. PMID 22984008
- [Result] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Result] Derdeyn CP, Chimowitz MI, Lynn MJ, Fiorella D, Turan TN, Janis LS, Montgomery J, Nizam A, Lane BF, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Lynch JR, Zaidat OO, Rumboldt Z, Cloft HJ; Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis Trial Investigators. Aggressive medical treatment with or without stenting in high-risk patients with intracranial artery stenosis (SAMMPRIS): the final results of a randomised trial. Lancet. 2014 Jan 25;383(9914):333-41. doi: 10.1016/S0140-6736(13)62038-3. Epub 2013 Oct 26. PMID 24168957
- [Derived] Siegler JE, Badillo Goicoechea E, Yaghi S, Morsi RZ, Arevalo A, Smith MM, Kothari S, Desai H, Sehgal N, Rana R, Kellogg CA, Jhaveri A, de Havenon A, Dunne T, Cameron K, Chaturvedi S, Ghannam M, Prabhakaran S, Coleman E, Brorson JR, Mehendale R, Kass-Hout T. Estimated Theoretical Benefit of Aggressive LDL Lowering in Patients With Symptomatic Intracranial Atherosclerosis. Neurology. 2025 Jul 8;105(1):e213768. doi: 10.1212/WNL.0000000000213768. Epub 2025 May 30. PMID 40446174
- [Derived] Wang T, Luo J, Li T, Almallouhi E, Gao P, Gong H, Zhang X, Wang J, Lu T, Yang Y, Yang R, Xing Z, Wang H, Derdeyn CP, Jiao L. Stenting versus medical treatment alone for symptomatic intracranial artery stenosis: a preplanned pooled individual patient data analysis. J Neurointerv Surg. 2025 Sep 12;17(10):1032-1039. doi: 10.1136/jnis-2024-022189. PMID 39147573
- [Derived] Yaghi S, Khatri P, de Havenon A, Yeatts S, Chang AD, Cutting S, Mac Grory B, Burton T, Jayaraman MV, McTaggart RA, Fiorella D, Derdeyn C, Zaidat OO, Dehkharghani S, Amin-Hanjani S, Furie K, Prahbakaran S, Liebeskind D. Peri-procedural stroke or death in stenting of symptomatic severe intracranial stenosis. J Neurointerv Surg. 2020 Apr;12(4):374-379. doi: 10.1136/neurintsurg-2019-015225. Epub 2019 Sep 4. PMID 31484697
- [Derived] Wabnitz AM, Derdeyn CP, Fiorella DJ, Lynn MJ, Cotsonis GA, Liebeskind DS, Waters MF, Lutsep H, Lopez-Cancio E, Turan TN, Montgomery J, Janis LS, Lane B, Chimowitz MI; SAMMPRIS Investigators. Hemodynamic Markers in the Anterior Circulation as Predictors of Recurrent Stroke in Patients With Intracranial Stenosis. Stroke. 2019 Jan;50(1):143-147. doi: 10.1161/STROKEAHA.118.020840. Epub 2018 Dec 11. PMID 30580705
- [Derived] Derdeyn CP, Fiorella D, Lynn MJ, Turan TN, Cotsonis GA, Lane BF, Montgomery J, Janis LS, Chimowitz MI; SAMMPRIS Investigators. Nonprocedural Symptomatic Infarction and In-Stent Restenosis After Intracranial Angioplasty and Stenting in the SAMMPRIS Trial (Stenting and Aggressive Medical Management for the Prevention of Recurrent Stroke in Intracranial Stenosis). Stroke. 2017 Jun;48(6):1501-1506. doi: 10.1161/STROKEAHA.116.014537. Epub 2017 Apr 28. PMID 28455321
- [Derived] Turan TN, Nizam A, Lynn MJ, Egan BM, Le NA, Lopes-Virella MF, Hermayer KL, Harrell J, Derdeyn CP, Fiorella D, Janis LS, Lane B, Montgomery J, Chimowitz MI. Relationship between risk factor control and vascular events in the SAMMPRIS trial. Neurology. 2017 Jan 24;88(4):379-385. doi: 10.1212/WNL.0000000000003534. Epub 2016 Dec 21. PMID 28003500
- [Derived] Waters MF, Hoh BL, Lynn MJ, Kwon HM, Turan TN, Derdeyn CP, Fiorella D, Khanna A, Sheehan TO, Lane BF, Janis S, Montgomery J, Chimowitz MI; Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) Trial Investigators. Factors Associated With Recurrent Ischemic Stroke in the Medical Group of the SAMMPRIS Trial. JAMA Neurol. 2016 Mar;73(3):308-15. doi: 10.1001/jamaneurol.2015.4315. PMID 26747792
- [Derived] Kwon HM, Lynn MJ, Turan TN, Derdeyn CP, Fiorella D, Lane BF, Montgomery J, Janis LS, Rumboldt Z, Chimowitz MI; SAMMPRIS Investigators. Frequency, Risk Factors, and Outcome of Coexistent Small Vessel Disease and Intracranial Arterial Stenosis: Results From the Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) Trial. JAMA Neurol. 2016 Jan;73(1):36-42. doi: 10.1001/jamaneurol.2015.3145. PMID 26618534
- [Derived] Lutsep HL, Lynn MJ, Cotsonis GA, Derdeyn CP, Turan TN, Fiorella D, Janis LS, Lane BF, Montgomery J, Chimowitz MI; SAMMPRIS Investigators. Does the Stenting Versus Aggressive Medical Therapy Trial Support Stenting for Subgroups With Intracranial Stenosis? Stroke. 2015 Nov;46(11):3282-4. doi: 10.1161/STROKEAHA.115.009846. Epub 2015 Sep 17. PMID 26382173
- [Derived] Chaturvedi S, Turan TN, Lynn MJ, Derdeyn CP, Fiorella D, Janis LS, Chimowitz MI; SAMMPRIS Trial Investigators. Do Patient Characteristics Explain the Differences in Outcome Between Medically Treated Patients in SAMMPRIS and WASID? Stroke. 2015 Sep;46(9):2562-7. doi: 10.1161/STROKEAHA.115.009656. Epub 2015 Aug 6. PMID 26251251
- [Derived] Lutsep HL, Barnwell SL, Larsen DT, Lynn MJ, Hong M, Turan TN, Derdeyn CP, Fiorella D, Janis LS, Chimowitz MI; SAMMPRIS Investigators. Outcome in patients previously on antithrombotic therapy in the SAMMPRIS trial: subgroup analysis. Stroke. 2015 Mar;46(3):775-9. doi: 10.1161/STROKEAHA.114.007752. Epub 2015 Jan 15. PMID 25593135
- See also: Clinical Alert — http://www.nlm.nih.gov/databases/alerts/intracranial_arterial_stenosis.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Medical Management Plus Stenting: intracranial angioplasty and stenting using the Gateway balloon and Wingspan self-expanding nitinol stent plus intensive medical therapy (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardiac indication, and aggressive risk factor management primarily targeting blood pressure < 140 / 90 mm Hg (< 130 / 80 if diabetic) and LDL < 70 mg / dl).
  intracranial angioplasty and stenting: intracranial angioplasty and stenting using the Gateway balloon and Wingspan self-expanding nitinol stent (or any future FDA approved iterations of the balloon, stent, or the delivery systems) plus intensive medical therapy (aspirin 325 mg / day for entire follow-up, clopidogrel 75mg per day for 90 days after enrollment unless cardiologist recommends continuing clopidogrel beyond 90 days for a cardia
Period: Overall Study
Arm/Group | Intensive Medical Management Plus Stenting | Intensive Medical Management Alone
Started | 224 | 227
Completed | 214 | 203
Not Completed | 10 | 24
Not completed — Lost to Follow-up | 7 | 11
Not completed — Withdrawal by Subject | 3 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Medical Management Plus Stenting | Intensive Medical Management Alone | Total
Number analyzed (Participants) | 224 | 227 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (10.7) | 59.5 (11.8) | 60.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 82 | 179
  Male | 127 | 145 | 272
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 55 | 49 | 104
  White | 160 | 162 | 322
  Other | 9 | 16 | 25
History of Hypertension [Number; unit: participants]
  Yes | 200 | 203 | 403
  No | 24 | 24 | 48
History of Lipid Disorder [Number; unit: participants]
  Yes | 195 | 202 | 397
  No | 29 | 25 | 54
Smoking [Number; unit: participants] — Based on the Physician-based Assessment and Counseling for Exercise (PACE) Smoking Score.
  The data value for smoking status was missing for 1 patient in the intensive medical management plus stenting group.
  participants
    Never | 90 | 78 | 168
    Previously | 79 | 80 | 159
    Currently | 54 | 69 | 123
Diabetes [Number; unit: participants] — A patient is considered diabetic at baseline if there is a history of diabetes or if the baseline hemoglobin A1c > 6.5%.
  participants
    Yes | 105 | 103 | 208
    No | 119 | 124 | 243
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 143.9 (20.6) | 146.8 (21.8) | 145.4 (21.3)
Low Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 96.2 (38.4) | 97.7 (36.6) | 97.0 (37.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (6.2) | 30.7 (6.3) | 30.5 (6.3)
History of Coronary Artery Disease [Number; unit: participants]
  Yes | 47 | 59 | 106
  No | 177 | 168 | 345
History of Stroke (Not Qualifying Event) [Number; unit: participants]
  Yes | 60 | 58 | 118
  No | 164 | 169 | 333
Qualifying Event [Number; unit: participants]
  Stroke | 142 | 152 | 294
  TIA | 82 | 75 | 157
On Antithrombotic Therapy at Qualifying Event [Number; unit: participants]
  Yes | 144 | 140 | 284
  No | 80 | 87 | 167
Time from Qualifying Event to Randomization [Median (Inter-Quartile Range); unit: days] | 7 [4 to 16] | 7 [4 to 19] | 7 [4 to 17.5]
Symptomatic Qualifying Artery [Number; unit: participants]
  Internal Carotid Artery | 45 | 49 | 94
  Middle Cerebral Artery | 92 | 105 | 197
  Vertebral Artery | 38 | 22 | 60
  Basilar Artery | 49 | 51 | 100
Percent Stenosis of Symptomatic Qualifying Artery [Mean (Standard Deviation); unit: % of the diameter the artery] — According to a reading of the cerebral angiogram by the site interventionist.
  % of the diameter the artery | 80 (7) | 81 (7) | 81 (7)

OUTCOME MEASURES:

1. Primary Outcome: Any Stroke or Death Within 30 Days of Enrollment or Any Revascularization Procedure OR an Ischemic Stroke in the Territory of the Symptomatic Intracranial Artery Beyond 30 Days After Enrollment.
Description: Any stroke (ischemic, parenchymal brain hemorrhage, subarachnoid or intraventricular hemorrhage) or death within 30 days after enrollment OR any stroke (ischemic, parenchymal brain hemorrhage, subarachnoid or intraventricular hemorrhage) or death within 30 days of any revascularization procedure of the qualifying symptomatic intracranial artery done during follow-up, OR an ischemic stroke in the territory of the symptomatic intracranial artery from day 31 after study entry to completion of follow-up.
Time Frame: Mean length of follow-up was 2.4 years
Population: All patients enrolled in the study were included in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | Intensive Medical Management Plus Stenting | Intensive Medical Management Alone
Number analyzed (Participants) | 224 | 227
participants | 52 | 34
Statistical Analysis 1: Comparison: Intensive Medical Management Plus Stenting vs Intensive Medical Management Alone; The statistical analysis was based on a comparison of the of the two treatment groups with respect to the time to a primary outcome using the logrank test; Test type: Superiority or Other; p = 0.0252, Log Rank

ADVERSE EVENTS:
Time Frame: Mean length of follow-up was 2.4 years
Description: The prespecified study outcomes were explicitly requested on the adverse event form. Any other adverse event was to be reported if it was either serious or related to a study intervention according to prespecified criteria and classified on the adverse event form using the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Arm/Group | Intensive Medical Management Plus Stenting | Intensive Medical Management Alone
Serious Adverse Events (participants affected / at risk) | 146/224 | 121/227
Other Adverse Events (participants affected / at risk) | 117/224 | 118/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Medical Management Plus Stenting (N=224) | Intensive Medical Management Alone (N=227)
Ischemic Stroke in the Territory of Qualifying Symptomatic Artery (Nervous system disorders) | 40 | 30
Ischemic Stroke Not in the Territory of the Qualifying Symptomatic Artery (Nervous system disorders) | 5 | 10
Symptomatic Intracranial Hemorrhage (Nervous system disorders) | 12 | 1
Intracranial Hematoma (Nervous system disorders) | 0 | 1
Transient Ischemic Attack / Cerebral Infarct with Temporary Signs (Nervous system disorders) | 30 | 29
Myocardial Infarction (Cardiac disorders) | 5 | 9
Systemic Hemorrhage (General disorders) | 15 | 8
Allergy / Immunology (Immune system disorders) | 3 | 0
Auditory / Ear (Ear and labyrinth disorders) | 1 | 1
Blood / Bone Marrow (Blood and lymphatic system disorders) | 4 | 3
Cardiac Arrhythmia (Cardiac disorders) | 13 | 7
Cardiac General (Cardiac disorders) | 14 | 18
Coagulation (Blood and lymphatic system disorders) | 0 | 1
Constitutional Symptoms (General disorders) | 2 | 2
Dermatology / Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Endocrine (Endocrine disorders) | 3 | 2
Gastrointestinal (Gastrointestinal disorders) | 13 | 12
Hepatobiliary / Pancreas (Hepatobiliary disorders) | 3 | 3
Infection (Infections and infestations) | 10 | 5
Lymphatics (Blood and lymphatic system disorders) | 1 | 0
Metabolic / Laaboratory (Metabolism and nutrition disorders) | 10 | 14
Musculoskeletal / Soft Tissue (Musculoskeletal and connective tissue disorders) | 8 | 6
Neurology (Nervous system disorders) | 26 | 19
Ocular / Visual (Eye disorders) | 3 | 5
Pain (General disorders) | 9 | 9
Pulmonary / Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Renal / Genitourinary (Renal and urinary disorders) | 10 | 5
Sexual / Reproductive (Reproductive system and breast disorders) | 2 | 1
Surgery / Intraoperative Injury (Surgical and medical procedures) | 4 | 3
Vascular (Vascular disorders) | 10 | 6
Asymptomatic Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Hemorrhage / Bleeding (Blood and lymphatic system disorders) | 1 | 0
Death (General disorders) | 13 | 13
Pulmonary Embolus (Vascular disorders) | 0 | 2
Cerebral Venous Thrombosis (Vascular disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 2
Complications of Acute Ischemia of a Limb or Internal Organ (Vascular disorders) | 4 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Medical Management Plus Stenting (N=224) | Intensive Medical Management Alone (N=227)
Transient Ischemic Attack / Cerebral Infarct with Temporary Signs (Nervous system disorders) | 27 | 34
Systemic Hemorrhage (General disorders) | 29 | 24
Cardiac General (Cardiac disorders) | 39 | 35
Gastrointestinal (Gastrointestinal disorders) | 5 | 15
Metabolic / Laboratory (Metabolism and nutrition disorders) | 17 | 13
Musculoskeletal / Soft Tissue (Musculoskeletal and connective tissue disorders) | 21 | 9
Neurology (Nervous system disorders) | 25 | 25
Pain (General disorders) | 14 | 11
Pulmonary / Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No